CLINICAL TRIAL: NCT01867294
Title: A Two-Part, Phase II Randomized Trial to Explore Topical Spironolactone to Prevent/Attenuate Rash From Epidermal Growth Factor Receptor Inhibitors (Panitumumab and Cetuximab) in Advanced Cancer Patients
Brief Title: Spironolactone in Preventing Rash in Patients With Advanced Cancer Receiving Panitumumab and Cetuximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC09C8; NCI-2012-01275 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RC09C8 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH); NCT02257086 (obsolete NCT alias)
Record Dates: First submitted 2012-08-27; First posted 2013-06-04 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2018-01

CONDITIONS: Advanced Malignant Neoplasm; Dermatologic Complication
MeSH Terms: interventions — Doxycycline; Spironolactone; Acetates; Sunscreening Agents; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm I (Study I) (Experimental): Patients apply spironolactone topically to face BID for 4 weeks.
  Interventions: Other: Questionnaire Administration; Drug: Spironolactone
- Arm I (Study II) (Experimental): Patients apply spironolactone topically to face and body BID for 4 weeks.
  Interventions: Other: Questionnaire Administration; Drug: Spironolactone
- Arm II (Study I) (Placebo Comparator): Patients apply placebo topically to face BID for 4 weeks.
  Interventions: Other: Placebo; Other: Questionnaire Administration
- Arm II (Study II) (Active Comparator): Patients receive modified preemptive therapy regimen consisting of skin moisturizer topically BID, sunscreen topically as needed, hydrocortisone topically QD, and doxycycline PO BID for 4 weeks.
  Interventions: Drug: Doxycycline; Procedure: Management of Therapy Complications; Other: Questionnaire Administration; Drug: Sunscreen; Drug: Therapeutic Hydrocortisone

INTERVENTIONS:
Drug: Doxycycline — Given PO
  Other Names: Doxycycline Monohydrate
  Arms: Arm II (Study II)
Procedure: Management of Therapy Complications — Moisturizer given topically
  Arms: Arm II (Study II)
Other: Placebo — Given topically
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (Study I)
Other: Questionnaire Administration — Ancillary studies
Drug: Spironolactone — Given topically
  Other Names: 17-Hydroxy-7alpha-mercapto-3-oxo-17alpha-pregn-4-ene-21-carboxylic Acid, gamma Lactone, Acetate; Aldactone; SC 9420; SPL
  Arms: Arm I (Study I); Arm I (Study II)
Drug: Sunscreen — Given topically
  Other Names: Sunblock
  Arms: Arm II (Study II)
Drug: Therapeutic Hydrocortisone — Given topically
  Other Names: Aeroseb-HC; Barseb HC; Barseb-HC; Cetacort; Cort-Dome; Cortef; Cortenema; Cortifan; Cortisol; Cortispray; Cortril; Dermacort; Domolene; Eldecort; Hautosone; Heb-Cort; hydrocortisone; Hydrocortone; Hytone; Komed-HC; Nutracort; Proctocort; Rectoid
  Arms: Arm II (Study II)

SUMMARY:
This randomized phase II trial studies how well giving spironolactone works in preventing rash in patients with cancer that has spread to other places in the body and are receiving panitumumab and cetuximab. Spironolactone may prevent endothelial growth factor receptor (EGFR) inhibitor-induced skin rash.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine feasibility of the administration of topical spironolactone versus placebo in this patient population. (Study I) II. To further explore the efficacy of the topical spironolactone to prevent/attenuate rash from EGFR inhibitors. (Study II)

SECONDARY OBJECTIVES:

I. To explore efficacy of the spironolactone versus placebo. (Study I) II. To describe the efficacy of a Modified Preemptive Therapy Regimen intervention. (Study II) III. To explore the adverse event profile of spironolactone and the Modified Preemptive Therapy Regimen intervention. (Study II) IV. To explore patient reported outcomes of patients using spironolactone and a Modified Preemptive Therapy Regimen intervention. (Study II) V. To explore long term (8 week) effect of the 4 week treatment of spironolactone and a Modified Preemptive Therapy Regimen intervention on EFGR induced rash. (Study II)

OUTLINE:

STUDY I: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients apply spironolactone topically to face twice daily (BID) for 4 weeks.

ARM II: Patients apply placebo topically to face BID for 4 weeks.

STUDY II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients apply spironolactone topically to face and body BID for 4 weeks

ARM II: Patients undergo modified preemptive therapy regimen consisting of skin moisturizer topically BID, sunscreen topically before going outside, hydrocortisone topically once daily (QD), and doxycycline orally (PO) BID for 4 weeks.

After completion of study, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to start panitumumab or cetuximab; patients must not have been on the EGFR agent prior to randomization
* Ability to reliably apply topical spironolactone/placebo twice a day to the face
* Ability to complete questionnaire(s) by themselves or with assistance
* For study 2 only, patients must be willing to avoid sun exposure for one month from registration
* Creatinine =< 1.5 x upper limit of normal (UNL)
* For Study 2 only, ability to apply topical creams to the entire face and body

Exclusion Criteria:

* Prior allergic reaction or severe intolerance to spironolactone
* Any rash at the time of randomization
* Cutaneous metastases
* Any other disorder that may predispose to hyperkalemia in the opinion of the treating oncologist
* Use of topical corticosteroids at the time of study or their anticipated use in the next 8 weeks; (it is acknowledged that patients may be starting these agents pre-emptively as part of this protocol)
* For study 2 only, previous intolerance of sunscreen or any of the other components of the Modified Preemptive Therapy Regimen (a moisturizer or oral doxycycline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-08-31 (Actual); Primary Completion 2014-05-09 (Actual); Study Completion 2014-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, Principal Investigator — Academic and Community Cancer Research United
Locations (5):
- United States (5):
  - Carle Cancer Center, Urbana, Illinois
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Marshfield Clinic, Marshfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study II was never opened due to the accrual rate in Study I.
Groups:
- Study I: Spironolactone: Patients apply spironolactone topically to face BID for 4 weeks.
- Study I: Placebo: Patients apply placebo topically to face BID for 4 weeks.
- Study II: Spironolactone: Patients apply spironolactone topically to face and body BID for 4 weeks.
- Study II: Modified Therapy: Patients receive modified preemptive therapy regimen consisting of skin moisturizer topically BID, sunscreen topically as needed, hydrocortisone topically QD, and doxycycline PO BID for 4 weeks.
Period: Overall Study
Arm/Group | Study I: Spironolactone | Study I: Placebo | Study II: Spironolactone | Study II: Modified Therapy
Started | 9 | 10 | 0 | 0
Completed | 8 | 9 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients that were treated and eligible for endpoint analysis were include in baseline characteristics. One patient from Study I: Spironolactone and one from Study I: Placebo withdrew from study participation prior to receiving any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Study I: Spironolactone | Study I: Placebo | Study II: Spironolactone | Study II: Modified Therapy | Total
Number analyzed (Participants) | 8 | 9 | 0 | 0 | 17
Age, Continuous [Median (Full Range); unit: years] | 65.0 [55.0 to 77.0] | 60.6 [39.0 to 82.0] |  |  | 62.6 [39 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 |  |  | 4
  Male | 6 | 7 |  |  | 13
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 |  |  | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting a Grade 2+ Adverse Event Attributed to Spironolactone (Study I)
Description: Adverse events were collected at the end of one 4-week cycle and one 4-week observation period according to the Common Terminology Criteria for Adverse Events (CTCAE) CTEP Version 4.0. The number of patients reporting a grade 2+ adverse event attributed to spironolactone is reported here.
Time Frame: At 8 weeks
Population: All patients that began study treatment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Study I: Spironolactone | Study I: Placebo | Study II: Spironolactone | Study II: Modified Therapy
Number analyzed (Participants) | 8 | 9 | 0 | 0
Participants | 0 | 0 |  |

2. Primary Outcome: Incidence of Truncal/Extremity Rash of Any Grade in Patients in the Spironolactone Arm (Study I)
Description: Adverse events were collected at the end of each 4-week cycle according to the Common Terminology Criteria for Adverse Events (CTCAE) CTEP Version 4.0. The number of patients reporting a truncal/extremity adverse event is reported here. The treatment will be considered feasible if at least 50% of patients in the spironolactone arm develop a truncal/extremity rash of any grade at the end of 4 weeks.
Time Frame: At 4 weeks
Population: All patients that began protocol treatment are included in this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Study I: Spironolactone | Study I: Placebo | Study II: Spironolactone | Study II: Modified Therapy
Number analyzed (Participants) | 8 | 9 | 0 | 0
Participants | 6 | 6 |  |

3. Primary Outcome: Percentage of Patients in the Spironolactone Arm Who Complete the 4-week Study Intervention (Study I)
Description: The number of patients able to complete the 4-week study intervention and the 4-week observation period are reported.
Time Frame: At 4 weeks
Population: All patients that began Study I treatment were included in this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Study I: Spironolactone | Study I: Placebo | Study II: Spironolactone | Study II: Modified Therapy
Number analyzed (Participants) | 8 | 0 | 0 | 0
Participants | 4 | 0 |  |

4. Primary Outcome: Efficacy of the Spironolactone Treatment to Prevent/Attenuate Rash From EGFR Inhibitors in This Patient Population Defined as Absence of Any Grade 2 or Worse Rash (Study II)
Description: The primary analysis will be descriptive in nature, and will involve an intent-to-treat analysis at the end of week 4. Patients will be categorized dichotomously according to healthcare provider reported grade 2 or worse rash. The absence of any grade 2 or worse rash will be a success and the existence of any such rash will be a failure. Patients who do not complete the 4 week treatment will be considered a failure. Point estimates and 95% confidence limits will be calculated.
Time Frame: At 4 weeks
Population: Study II was not conducted.
Arm/Group | Study I: Spironolactone | Study I: Placebo | Study II: Spironolactone | Study II: Modified Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Efficacy of Spironolactone and Placebo Measured by the Use of the Brief Pictorial Rash Incidence Questionnaire (Study I)
Description: Patients will be dichotomously categorized as a success if no rash is reported and a failure if rash exists at the end of 4 weeks. The number of patients that successfully completed 4 weeks of treatment and reported no rash on the Brief Pictorial Rash Incidence Questionnaire are reported.
Time Frame: At 4 weeks
Population: All patients that began study treatment are included in this analysis.
Measure: Number; unit: participants
Arm/Group | Study I: Spironolactone | Study I: Placebo | Study II: Spironolactone | Study II: Modified Therapy
Number analyzed (Participants) | 8 | 9 | 0 | 0
participants | 1 | 2 |  |

6. Secondary Outcome: Efficacy of the Modified Preemptive Therapy Regimen, Calculated and Analyzed Analogously to the Efficacy of the Spironolactone (Study II)
Description: All secondary endpoints will be reported descriptively using frequency statistics and single sample t-tests. Outcomes with respect to baseline covariates will also be explored.
Time Frame: At 4 weeks
Population: Study II was not conducted.
Arm/Group | Study I: Spironolactone | Study I: Placebo | Study II: Spironolactone | Study II: Modified Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Efficacy of the Spironolactone Treatment to Prevent/Attenuate Rash From EGFR Inhibitors in This Patient Population Defined as Absence of Any Grade 2 or Worse Rash (Study II)
Description: This analysis will be descriptive in nature, and will involve an intent-to-treat analysis at the end of week 8. Patients will be categorized dichotomously according to healthcare provider reported grade 2 or worse rash. The absence of any grade 2 or worse rash will be a success and the existence of any such rash will be a failure. Patients who do not complete the 8 week treatment will be considered a failure. Point estimates and 95% confidence limits will be calculated.
Time Frame: At 8 weeks
Population: Study II was not conducted.
Arm/Group | Study I: Spironolactone | Study I: Placebo | Study II: Spironolactone | Study II: Modified Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Incidence of Healthcare Provider Reported Adverse Events (Study II)
Description: as for outcome 6
Time Frame: At 8 weeks
Population: Study II was not conducted.
Arm/Group | Study I: Spironolactone | Study I: Placebo | Study II: Spironolactone | Study II: Modified Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Patient Reported Outcomes as Measured by the Change From Baseline in the SKINDEX-16 Total Score (Study II)
Description: Total scores from the SKINDEX-16 will be compared from baseline to week 4. Comparisons between treatment arms will be made by t-tests.
Time Frame: At 4 weeks
Population: Study II was not conducted.
Arm/Group | Study I: Spironolactone | Study I: Placebo | Study II: Spironolactone | Study II: Modified Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed after one 4 week cycle, and after one 4-week observation prior for a maximum of up to 8 weeks.
Description: Adverse events were assessed after one 4 week cycle, and after one 4-week observation prior for a maximum of up to 8 weeks.
Groups:
- Study I: Spironolactone: .Patients apply spironolactone topically to face BID for 4 weeks.
Arm/Group | Study I: Placebo | Study I: Spironolactone
All-Cause Mortality (participants affected / at risk) | 2/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/9 | 2/8
Other Adverse Events (participants affected / at risk) | 8/9 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study I: Placebo (N=9) | Study I: Spironolactone (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study I: Placebo (N=9) | Study I: Spironolactone (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8) | 5 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (9) | 6 (10)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No